CLINICAL TRIAL: NCT01519128
Title: A Phase I, Open Label, Randomized, Crossover Trial in Healthy Subjects to Investigate the Effect of Steady-state TMC278 on the Pharmacokinetics of a Single Dose of Digoxin
Brief Title: A Study to Investigate the Effect of Steady-State TMC278 on the Pharmacokinetics of a Single Dose of Digoxin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen R&D Ireland (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR100750; TMC278IFD1001 (Other: Janssen R&D Ireland); 2011-004159-38 (EudraCT Number)
Record Dates: First submitted 2011-12-27; First posted 2012-01-26 (Estimated); Last update posted 2013-03-04 (Estimated); Status verified 2013-03

CONDITIONS: Healthy
Keywords: Healthy; TMC278; TMC278IFD1001; Human immunodeficiency virus - type 1; Pharmacokinetics; Digoxin
MeSH Terms: conditions — Acquired Immunodeficiency Syndrome | interventions — Digoxin; Rilpivirine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Treatment sequence AB (Experimental): In Treatment A, digoxin 0.5 mg (single oral dose) will be administered on Day 1. In Treatment B, TMC278 at 25 mg, once daily will be administered for 16 days, with digoxin 0.5 mg (single oral dose) administered in the morning on Day 11.
  Interventions: Drug: Treatment A: Digoxin; Drug: Treatment B: TMC278
- Treatment sequence BA (Experimental): In Treatment B, TMC278 at 25 mg, once daily will be administered for 16 days, with digoxin 0.5 mg (single oral dose) administered in the morning on Day 11. In Treatment A, digoxin 0.5 mg (single oral dose) will be administered on Day 1.
  Interventions: Drug: Treatment A: Digoxin; Drug: Treatment B: TMC278

INTERVENTIONS:
Drug: Treatment A: Digoxin — Type=exact number, unit=mg, number=0.5, form=tablet, route=oral. Digoxin administered on Day 1.
  Other Names: Digoxin
Drug: Treatment B: TMC278 — Type=exact number, unit=mg, number=25, form=tablet, route=oral. TMC278 administered for 16 days, with digoxin administered in the morning on Day 11.
  Other Names: TMC278

SUMMARY:
The purpose of this study is to investigate the effect of steady-state (constant concentration of medication in the blood) TMC278 on the single dose pharmacokinetics (what the body does to the medication) of digoxin.

DETAILED DESCRIPTION:
This is an open-label (all people know the identity of the intervention), randomized (the study medication is assigned by chance), crossover (method used to switch patients from one treatment arm to another in a clinical study) study to investigate the effect of steady-state TMC278 on the single dose pharmacokinetics of digoxin. The study consists of 3 phases, including screening phase, treatment phase, and follow-up phase. After the screening phase, participants will be randomized to one of 2 treatment sequences consisting of Treatments A and B, ie, Sequence AB (11 participants), and Sequence BA (11 participants). Treatment phase includes, Treatment A: digoxin 0.5 mg (single oral dose), and Treatment B: TMC278 25 mg once daily with digoxin 0.5 mg (single oral dose). The 2 consecutive sequences will be separated by a washout period (period when receiving no treatment) of at least 14 days. Safety evaluations for adverse events, clinical laboratory tests, electrocardiograms, cardiac telemetry, vital signs, physical examination, alcohol breath test, and specific toxicities will be monitored throughout the study.The study duration for treatment phase will be at least 26 days.

ELIGIBILITY:
Inclusion Criteria:

* Women must be postmenopausal for at least 2 years, or be surgically sterile
* Men must agree to use a highly effective method of birth control and to not donate sperm during the study and for 3 months after receiving the last dose of study medication

Exclusion Criteria:

* A positive HIV-1 or HIV-2 test at screening
* Hepatitis A, B or C infection at screening
* History of clinically relevant heart rhythm disturbances
* History of idiopathic hypertrophic subaortic stenosis, atrioventricular block, ventricular tachycardia/ventricular fibrillation or family history of sudden cardiac death

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2012-01; Primary Completion 2012-04 (Actual); Study Completion 2012-04 (Actual)

PRIMARY OUTCOMES:
Maximum plasma concentration (Cmax) of digoxin following single dose administration of digoxin co-administered with TMC278, compared to single dose administration of digoxin | Up to 46 Days
  Pharmacokinetic parameter Cmax of digoxin was measured following single dose administration of digoxin co-administered with TMC278, compared to single dose administration of digoxin.
Area under the plasma concentration versus time curve (AUC) of digoxin following single dose administration of digoxin co-administered with TMC278, compared to single dose administration of digoxin | Up to 46 Days
  Pharmacokinetic parameter AUC of digoxin was measured following single dose administration of digoxin co-administered with TMC278, compared to single dose administration of digoxin.

SECONDARY OUTCOMES:
Number of participants with adverse events | Up to 58 Days

CONTACTS AND LOCATIONS:
Overall Officials: Janssen R&D Ireland Clinical Trial, Study Director — Janssen R&D Ireland
Locations (1):
- Merksem, Belgium

REFERENCES:
- See also: A Phase I, open label, randomized, crossover trial in healthy subjects to investigate the effect of steady-state TMC278 on the pharmacokinetics of a single dose of digoxin. — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3415&filename=CR100750_CSR.pdf